CLINICAL TRIAL: NCT03283176
Title: Changes in Hematologic Profile, Vitamin B12 and Folic Acid Level in Cirrhotic Patients Received Sofosbuvir and Daclatasvir With or Without Ribavirin
Brief Title: Hematologic Profile, Vit. B12 and Folic Acid in Cirrhotics Received Sofosbuvir and Daclatasvir With or Without Ribavirin
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Shaaban Redwan Helal, Resident doctor at Tropical Medicine and Gastroenterology Department, Assiut University
Other Study IDs: Haematological Prof. in DAAs
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Liver Cirrhoses; Chronic Hepatitis c; Directly Acting Antivirals
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sofo-Dacla with Ribavirin: Chronic Hepatitis C related Liver Cirrhosis patients who will take sofosbuveir, Daclatasvir with Ribavirin
  Interventions: Diagnostic Test: Vitamin B12 and Folic Acid
- Sofo-Dacla without Ribavirin: Chronic Hepatitis C related Liver Cirrhosis patients who will take sofosbuveir, Daclatasvir without Ribavirin
  Interventions: Diagnostic Test: Vitamin B12 and Folic Acid

INTERVENTIONS:
Diagnostic Test: Vitamin B12 and Folic Acid — Vitamin B12 and Folic Acid measurement by ELISA technique

SUMMARY:
Use of Ribavirin could affect hematologic profile of the patients negatively. With advent of new antiviral therapy, the preexisting hematologic changes may alter or corrected after treatment. However, this point is still not properly studied.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection is a global health problem that affects 170 million people worldwide, and approximately 55% (95 million) of the infected population is in South East Asia and Western Pacific countries.

Hepatitis C virus (HCV) is considered one of the main causes of chronic hepatitis and also may be complicated by serious complications as liver cirrhosis, ascites and hepatocellular carcinoma. It is also, one of the leading indications for liver transplantation (LT) in adults around the world.

Abnormalities in hematological parameters are common in patients with cirrhosis. The pathogenesis of abnormal hematological indices (HIs) in cirrhosis is multifactorial and includes portal hypertension-induced sequestration, alterations in bone marrow stimulating factors, viral- and toxin-induced bone marrow suppression and consumption or loss. Abnormalities in HIs are associated with an increased risk of complications including bleeding and infection.

So, early recognition and early treatment of those patients with chronic HCV infection can modify its natural history. There are many factors affecting the outcome of HCV infection as viral, environmental and host factors, including immunologic and genetic susceptibilities.

Till 2011, the main lines of therapy were Interferon plus ribavirin for at least 48 weeks but these combinations was associated with low incidence of Sustained Virological Response (SVR). Now, there is era of Direct Acting Analogues that used for treatment of patients with chronic HCV infection and associated with high rate of SVR.

Daclatasvir is a first-in-class HCV NS5A replication complex inhibitor, and Sofosbuvir is a nucleotide analogue HCV NS5B polymerase inhibitor. Both have potent antiviral activity and broad genotypic coverage and are administered orally once daily.

ELIGIBILITY:
Inclusion Criteria:

* Patients known to have HCV-related liver cirrhosis and candidate for therapy with Sofosbuvir and Daclatasvir with or without Ribavirin

Exclusion Criteria:

* Chronic hepatitis due causes other than chronic HCV infection
* Coinfection with HIV or HBV infection
* Hepatocellular carcinoma
* Decompensated cirrhosis

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Fifty patients were diagnosed to have HCV-related liver cirrhosis and candidate for anti- HCV therapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Vitamin B12 | 1 year
  By ELISA Technique, in Pg/ml
Folic Acid | 1 year
  By ELISA technique, in Pg/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Shaban Redwan Helal, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghany MG, Strader DB, Thomas DL, Seeff LB; American Association for the Study of Liver Diseases. Diagnosis, management, and treatment of hepatitis C: an update. Hepatology. 2009 Apr;49(4):1335-74. doi: 10.1002/hep.22759. No abstract available. PMID 19330875
- [Background] Promrat K, McDermott DH, Gonzalez CM, Kleiner DE, Koziol DE, Lessie M, Merrell M, Soza A, Heller T, Ghany M, Park Y, Alter HJ, Hoofnagle JH, Murphy PM, Liang TJ. Associations of chemokine system polymorphisms with clinical outcomes and treatment responses of chronic hepatitis C. Gastroenterology. 2003 Feb;124(2):352-60. doi: 10.1053/gast.2003.50061. PMID 12557141
- [Background] Lam AM, Espiritu C, Bansal S, Micolochick Steuer HM, Niu C, Zennou V, Keilman M, Zhu Y, Lan S, Otto MJ, Furman PA. Genotype and subtype profiling of PSI-7977 as a nucleotide inhibitor of hepatitis C virus. Antimicrob Agents Chemother. 2012 Jun;56(6):3359-68. doi: 10.1128/AAC.00054-12. Epub 2012 Mar 19. PMID 22430955
- [Background] Ampuero J, Romero-Gomez M, Reddy KR. Review article: HCV genotype 3 - the new treatment challenge. Aliment Pharmacol Ther. 2014 Apr;39(7):686-98. doi: 10.1111/apt.12646. PMID 24612116
- [Background] Qamar AA, Grace ND. Abnormal hematological indices in cirrhosis. Can J Gastroenterol. 2009 Jun;23(6):441-5. doi: 10.1155/2009/591317. PMID 19543577